CLINICAL TRIAL: NCT03640533
Title: The Efficacy of the Nanit-Insights App in Improving Infant Sleep: A Randomized Controlled Trial
Brief Title: The Efficacy of the Nanit-Insights App in Improving Infant Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical probelms led to inadequate randomization, and thus the project was terminated.
Sponsor: Tel Aviv University (Other)
Collaborators: Flinders University (Other); UdiSense Inc. (Unknown)
Responsible Party: Principal Investigator, Michal Kahn, Post-doctoral fellow, Children's Sleep Laboratory, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Insights
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Infant Sleep Problems

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanit-Insights intervention group (Experimental): Nanit-Insights is an app-based intervention that provides parents with personalized sleep recommendations, based on their infant's developmental stage and weekly sleep data.
  Interventions: Behavioral: Nanit-Insights
- Nanit-monitor control group (No Intervention): Participants in the control group will be given the same monitoring device, that will serve in this group as a baby-monitor only, without providing sleep recommendations to parents.

INTERVENTIONS:
Behavioral: Nanit-Insights — Nanit-Insights is an app-based intervention that provides personalized sleep tips to parents.
  Arms: Nanit-Insights intervention group

SUMMARY:
The proposed study aims to examine the effectiveness of Nanit-Insights, an app-based intervention for parents who wish to improve their infant's sleep.

DETAILED DESCRIPTION:
The proposed study aims to examine the effectiveness of Nanit-Insights, an app-based intervention for parents who wish to improve their infant's sleep. The intervention provides parents with daily sleep metrics as well as personalized sleep recommendations, based on their infant's developmental stage and weekly sleep data.

Participants will be parents of 5-7 month-old infants, randomized into one of two groups: (1) the intervention group, which will include users who have purchased the baby monitor without subscribing to Nanit Insights and are then offered a six month subscription to Nanit-Insights when their baby is 5-7 months of age; and (2) the control group, which will include users of the baby monitor, who have not subscribed to Nanit-Insights.

Each group will include approximately 150 families.

Sleep will be assessed at baseline and 3- and 6-months following the beginning of the intervention. Computer vision technology will be used to assess infant sleep, as well as parental adherence to the intervention, allowing us to determine whether adherence mediates sleep benefits.

The results of this study are expected to evaluate the effectiveness of a low-cost, app-based intervention for infant sleep problems. Furthermore, the results may broaden the understanding of the mediating role of parent adherence in such interventions.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 5-7 months
* Presence of a moderate to severe sleep problem at baseline
* Sleeping arrangement in which the infant sleeps in a crib at night

Exclusion Criteria:

-

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent-reported infant sleep quality at 3 and 6 months follow-up as assessed using the Extended Brief Infant Sleep Questionnaire | Infant sleep quality will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in parent-reported sleep quality at 3 and 6 months follow-up using the Extended Brief Infant Sleep Questionnaire. Items in this questionnaire are either open-ended or reported on a 5-point scale, with 1=poor sleep quality and 5=very good sleep quality.
Change from baseline in infant sleep efficacy at 3 and 6 months follow-up: Videosomnography | Infant sleep efficacy will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of sleep efficacy at 3 and 6 months follow-up. infant sleep will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm. Sleep efficacy will be provided using the algorithm.

SECONDARY OUTCOMES:
Change from baseline in parent sleep quality as assessed using the Pittsburgh Sleep Quality Index at 3 and 6 month follow ups. | Parent sleep quality will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in parent-reported sleep quality using the Pittsburgh Sleep Quality Index (PSQI) at 3 and 6 month follow ups. The PSQI is comprised of 10 questions, from which the following subscales are generated: sleep latency, sleep duration, sleep disturbances, and daytime-dysfunction. Items are open-ended or rated on a 4-point scale, and higher scores represent poorer sleep.
Change from baseline in parent mood as assessed using the Clinically Useful Depression Outcome Scale at 3 and 6 month follow ups. | Parent mood will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in parent-reported mood using the Clinically Useful Depression Outcome Scale (CUDOS) at 3 and 6 month follow ups. Each of the 18 items in the CUDOS is rated on a 5-point scale, with higher ratings indicating poorer mood. Ratings on all items are summed to create a total score.
Change from baseline in infant sleep onset latency at 3 and 6 months follow-up: Videosomnography | Infant sleep onset latency will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of sleep onset latency at 3 and 6 months follow-up. Infant sleep will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm.
Change from baseline in infant sleep duration at 3 and 6 months follow-up: Videosomnography | Infant sleep duration will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of sleep duration at 3 and 6 months follow-up. Infant sleep will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm.
Change from baseline in infant number of night-wakings at 3 and 6 months follow-up: Videosomnography | Infant number of night-wakings will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of number of night-wakings at 3 and 6 months follow-up. Infant sleep will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm.
Change from baseline in infant time out of bed at 3 and 6 months follow-up: Videosomnography | Infant time out of bed will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of number of time out of bed at 3 and 6 months follow-up. Infant sleep will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm.
Change from baseline in parental "nightly visits" at 3 and 6 months follow-up: Videosomnography | Infant time out of bed will be assessed at baseline, and at 3- and 6-month follow-ups.
  Change from baseline in videosomnography metric of parental "nightly visits" to the crib at 3 and 6 months follow-up. Parental visits to the infant in the crib will be assessed for 10 consecutive nights using the Nanit videosomnography camera and algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kahn, PhD, Study Director — Tel Aviv University; Michael Gradisar, PhD, Principal Investigator — Flinders University
Locations (1):
- Nanit, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be encrypted, to ensure privacy of participants. It will be shared with investigators of the present study only.